CLINICAL TRIAL: NCT06612749
Title: Assessing the Impact of Integrative Medicine on Anxiety and Wellbeing of Healthcare Providers Exposed Directly or Indirectly to Terror, Trauma or War
Brief Title: Assessing the Impact of Integrative Medicine on Anxiety and Wellbeing of Healthcare Providers Exposed to Terror or War
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Director, Integrative Medicine Program, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15102023
Record Dates: First submitted 2024-08-25; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Quality of Life
Keywords: Resilience; Integrative medicine; Healthcare providers; Acupuncture
MeSH Terms: interventions — Acupuncture Therapy; Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative medicine intervention (Experimental): Healthcare providers were treated for 30 minutes with integrative medicine based on manual and mind-body modalities
  Interventions: Other: Integrative medicine including manual and/or mind-body treatments

INTERVENTIONS:
Other: Integrative medicine including manual and/or mind-body treatments — Referred HCPs are recommended a multi-modal IM program, include at least one of the following: acupuncture; manual-movement therapies (e.g., acupressure, Anthroposophic medicine touch therapies, reflexology, Qi Gong, and Feldenkrais method); and mind-body medicine (e.g., relaxation and breathing techniques).
  Other Names: Acupuncture; Relaxation; Acupressure

SUMMARY:
The study assesses integrative medicine intervention effects on healthcare providers' quality-of-life during wartime.

DETAILED DESCRIPTION:
The study is prospective, non-randomized and non-controlled, and taking place at the Carmel Medical Center in Haifa, northern Israel, from October 2023. The study was launched in proximity with the outbreak of the October 2023 war in the Middle East. As this timing was and is still regarded in Israel as an emergency life-threatening situation and considering the research limitation to healthcare providers only, the Carmel Medical Center Institutional Review Board has exempted the study from requiring written consent from participants, after reviewing the study protocol. However, Participation in the study was voluntary, and no incentive, financial or other was offered.

The hospital administration and department refer healthcare providers (HCPs) to integrative medicine intervention those if reporting emotional, physical, or other QoL concerns directly or indirectly related to the current conflict in Israel. The IM intervention entails a 30-minute treatment session, with an additional 10 minutes allocated for both pre- and post- treatment assessment. IM treatments are individually tailored to the HCP's QoL-related concerns, taking into consideration their willingness to undergo the recommended modalities. In all cases, a multi-modal IM program is recommended, which includes at least one of the following: acupuncture; manual-movement therapies (e.g., acupressure, Anthroposophic medicine touch therapies, reflexology, Qi Gong, and Feldenkrais method); and mind-body medicine (e.g., relaxation and breathing techniques). During these treatments participants are asked to lay on a treatment bed, with relaxed non-paced breathing throughout the session. The IM treatments are provided by IM-trained therapists who work in an integrative oncology setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers reporting war-related concerns affecting their quality of life

Exclusion Criteria:

* Healthcare providers with no quality-of-life related concerns they attribute to the war r

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessing HCPs QoL-related concerns using the Measure Yourself Concerns and Wellbeing (MYCAW). | Before and immediately following the IO intervention; and at 24-48 hours post-treatment.
  The MYCAW asks patients to list their two most significant concerns and general feeling of wellbeing (from 0, "doesn't bother me at all"; to 6, "bothers me greatly"). At post-treatment, the HCPs are asked to re-score the two original leading concerns and general well-being, followed by two open-ended questions about "Other things affecting your health"; and "What has been most important for you?" with respect to the IM treatments they had received. In the post-intervention narratives, HCPs are asked to describe the most important aspects of their treatment. HCP narratives are considered as free-text narratives, which may be qualitatively analyzed using ATLAS.Ti software for systematic coding, to identify clusters of emotional-spiritual keywords (ESKs), such as "calming", "release", "relaxation" and "disengagement".
Assessment of objective physiological changes during the intervention | During the 30 minutes intervention
  Assessment of objective physiological changes during the 30-minute intervention are conducted using chest-lead electrocardiogram monitoring autonomic heart rate variability (HRV) throughout the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben-Arye E, Gressel O, Samuels N, Stein N, Eden A, Vagedes J, Kassem S. Complementary and integrative medicine intervention in front-line COVID-19 clinicians. BMJ Support Palliat Care. 2022 Apr 5:bmjspcare-2021-003333. doi: 10.1136/bmjspcare-2021-003333. Online ahead of print. PMID 35383045
- [Background] Vagedes J, Kassem S, Gressel O, Samuels N, Eden A, Ben-Arye E. Parasympathetic Versus Sympathetic Changes in Heart Rate Variability After a Multimodal Integrative Medicine Intervention for Frontline COVID-19 Personnel. Psychosom Med. 2023 Jan 1;85(1):53-60. doi: 10.1097/PSY.0000000000001153. Epub 2022 Nov 9. PMID 36346679
- [Derived] Kassem S, Vagedes J, Gressel O, Samuels N, Elias S, Ben-Arye E. Spirit and Sense: Autonomic Response to Integrative Medicine Intervention for Health Care Personnel During Wartime. Biopsychosoc Sci Med. 2025 Jul-Aug 01;87(6):380-387. doi: 10.1097/PSY.0000000000001402. Epub 2025 Jun 11. PMID 40511976